CLINICAL TRIAL: NCT06995703
Title: Increasing Screening for Cancer Using EHR-Nudges, A Replication Trial
Brief Title: Increasing Screening for Cancer Using EHR-Nudges Replication
Acronym: I-SCREEN Rep
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Amol Navathe, Professor of Health Policy and Medicine, Abramson Cancer Center at Penn Medicine
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Health Services Research
Other Study IDs: UPCC 03025; R33AG068947 (NIH)
Record Dates: First submitted 2025-05-21; First posted 2025-05-29 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Breast Cancer
Keywords: Screening; Mammogram; Behavioral Economics; Prevention
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: In a 2x2 factorial design, eligible patients will be randomized in a 1:1 ratio on two factors: 1) receive a pre-visit text message (patient nudge) and Smart Data Element (SDE) message in the EHR (clinician nudge) or no pre-visit text and SDE message; and 2) receive post-visit text messaging or no post-visit text messaging.
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Pre-Visit Text Message/Smart Data Element Only (Experimental): Patients randomized to this arm will receive the pre-visit text message and Smart Data Element nudges.
  Interventions: Behavioral: Pre-Visit Patient Text Message; Behavioral: Smart Data Element (SDE)
- Pre-Visit Text Message/Smart Data Element + Post-Visit Text Message (Experimental): Patients randomized to this arm will be eligible to receive both the pre- and post-visit text messages and the Smart Data Element nudges.
  Interventions: Behavioral: Pre-Visit Patient Text Message; Behavioral: Post-Visit Patient Text Messages; Behavioral: Smart Data Element (SDE)
- Post-Visit Text Message Only (Experimental): Patients randomized to this arm will be eligible to receive the post-visit text message nudges.
  Interventions: Behavioral: Post-Visit Patient Text Messages
- Standard of Care (No Intervention): Patients randomized to the standard of care arm will receive no nudge interventions.

INTERVENTIONS:
Behavioral: Pre-Visit Patient Text Message — Patients will be sent a text message reminder 1 day prior to their scheduled primary care visit. This message will remind them of their upcoming appointment, highlight that they may be overdue for their mammogram, and encourage them to speak with their provider or schedule now by using the provided online scheduling link or phone number. Patients who do not have a cell phone number listed in the EHR will receive automated voice recording (AVR).
  Arms: Pre-Visit Text Message/Smart Data Element + Post-Visit Text Message; Pre-Visit Text Message/Smart Data Element Only
Behavioral: Post-Visit Patient Text Messages — Patients will be sent text message reminders 4 days and 14 days after their completed primary care visit if they have not yet scheduled or completed their screening mammogram. The message delivered at 4 days post-visit will remind the patient to schedule and that appointments are available for them. The message delivered at 14-days post-visit will again encourage the patient to schedule their mammogram, if one has not already been scheduled or completed. Both messages will include a scheduling phone number and link to self-schedule online. Patients who do not have a cell phone number listed in the EHR will receive automated voice recording (AVR).
  Arms: Post-Visit Text Message Only; Pre-Visit Text Message/Smart Data Element + Post-Visit Text Message
Behavioral: Smart Data Element (SDE) — The clinician-facing Smart Data Element (SDE) in the EHR will be visible to the provider and care team during the visit encounter. The SDE will display as a section in pre-charting, check-in, and rooming and will notify the clinician and care team that a pre-visit communication was sent to the patient regarding scheduling an overdue mammogram and including results from prior work that show that patients are more likely to complete their screening if they receive an order and recommendation from their provider.
  Arms: Pre-Visit Text Message/Smart Data Element + Post-Visit Text Message; Pre-Visit Text Message/Smart Data Element Only

SUMMARY:
In this study, personalized nudges to clinicians and patients will be evaluated to help increase breast cancer screening rates in accordance with USPSTF guidelines among women with a primary care visit. In partnership with Penn Medicine (Penn) and Case Western Reserve University-University Hospitals (UH), two complementary, concurrent 6-month, cluster randomized, pragmatic trials were conducted from December 2023 to October 2024. This trial will now replicate those interventions at Lancaster General Health (LGH), incorporating learnings from the primary trials while also adapting to align with existing health system protocols and policies. The patient nudge interventions include pre- and post-visit text message reminders to encourage the patient to schedule their mammogram, and the clinician nudge intervention includes a Smart Data Element message in the electronic health record (EHR) reminding the care team that the patient is overdue and that patients are more likely to complete their screening if recommended and ordered by their clinician.

DETAILED DESCRIPTION:
Cancer is a leading cause of mortality in the United States. While strong USPSTF guideline recommendations support appropriate screening for early detection and to avoid preventable deaths, breast cancer screening is often underutilized. Increasing breast cancer screening rates is challenging, in part, because it requires complementary decisions from clinicians (e.g., recommend and counsel patients about screening) and patients (e.g., to internalize risks and choose to complete screening). Presently, the lack of interventions directly targeting both clinicians' and patients' decision-making may underscore the relatively stagnant screening rates in the United States. There is a significant need to develop and scale low-cost interventions that increase breast cancer screening while simultaneously addressing the needs of high-risk patients and reducing disparities. Building upon prior work, the investigators propose to develop and test EHR-based clinician and patient nudges at a replication site (Lancaster General Health) to help increase screening mammography rates. The analyses will compare the effectiveness of clinician and patient nudges in the overall patient population and separately among high-risk patients to inform what methods are most effective for each of these populations.

ELIGIBILITY:
Inclusion Criteria:

All patients must meet the following criteria to be eligible:

1. Women between 40 and 74 years of age
2. A scheduled new or return (non-urgent/sick) primary care visit at one of the study practices at Lancaster General Health
3. Are overdue and eligible for a mammogram per Epic Health Maintenance
4. Does not have a future scheduled mammogram appointment

Patients meeting at least one of the following criteria will be considered high risk for screening non-completion:

1. Medicare Insurance
2. Medicaid Insurance
3. No EHR patient portal account
4. Zero log-ins to EHR patient portal in the previous year

Exclusion Criteria:

Patients will be excluded from the study if they:

1. Have a history of bilateral mastectomy, breast cancer, or metastatic cancer
2. Have a mammogram exclusion modifier in Health Maintenance
3. Have no phone number (home or mobile) listed in their chart

Ages: 40 Years to 74 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7920 (Estimated)
Dates: Start 2025-06-02 (Actual); Primary Completion 2026-03-02 (Estimated); Study Completion 2026-06-02 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients who complete a screening mammogram within 3 months after the visit | 3 months
  The primary outcome is screening mammogram completion within 3 months after the first eligible primary care visit.

SECONDARY OUTCOMES:
Proportion of patients who complete a screening mammogram within 6 months after the visit | 6 months
  The secondary outcome is screening mammogram completion within 6 months after the first eligible primary care visit.

OTHER OUTCOMES:
Difference in screening rates between high and low risk subgroups within 3 months after the visit | 3 months
  We will compare the difference in screening rates between the high and low risk subgroups amongst patients who were randomized to receive at least one type of nudge versus patients who were randomized to standard of care.

CONTACTS AND LOCATIONS:
Overall Officials: Amol Navathe, MD, PhD, Principal Investigator — University of Pennsylvania
Locations (1):
- Lancaster General Health, Lancaster, Pennsylvania, United States